CLINICAL TRIAL: NCT01289496
Title: Ribavirin Dose Optimization for the Treatment of Hepatitis C: A Pilot Study
Brief Title: Ribavirin Dose Optimization for the Treatment of Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Hoffmann-La Roche (Industry); Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25553; Control Number: 143155 (Other: Health Canada)
Record Dates: First submitted 2011-01-25; First posted 2011-02-03 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Hepatitis C
Keywords: Ribavirin; Pegasys; Hepatitis
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis | interventions — Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Peg-interferon alpha-2a, Ribavirin (Experimental): Adult patients with chronic hepatitis C and failure of prior treatment with peginterferon plus ribavirin(non-response or relapse).
  This is a pilot study with no control group.
  Interventions: Drug: Peg-interferon alpha-2a, Ribavirin

INTERVENTIONS:
Drug: Peg-interferon alpha-2a, Ribavirin — * 4 weeks RBV priming;
  * 24 or 48 weeks of Pegasys+Ribavirin (RBV) Treatment (depending on genotype);
  * 24 weeks Follow-Up
  Patients will receive PEGASYS® 180 µg in 0.5 mL (prefilled syringes) administered sc once weekly. Specific guidelines for adjusting the dose of PEGASYS® are provided in the product monograph.All PEGASYS® administrations will be via the sc route using sterile technique.
  Ribavirin 200 mg tablets
  Other Names: Peg-interféron alpha-2a (PEGASYS); Ribavirin (COPEGUS)

SUMMARY:
Patients for whom treatment with peginterferon plus ribavirin was unsuccessful represent a category of patients for whom there is currently no worthwhile therapeutic alternative.

Several studies have shown that there is a relation between plasma ribavirin concentrations and treatment response. Adequate ribavirin plasma concentrations, especially during the first 12 weeks of treatment, should be associated with a better chance of response to the treatment.

The strategy for this study will be to use a loading dose of ribavirin before beginning the treatment with peg-interferon, thereby allowing for optimal ribavirin concentrations to be reached, and possibly improving the effectiveness of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Chronic hepatitis C and failure of prior treatment with peginterferon plus ribavirin (non-response: HCV-RNA decreased less than 2 logs after 3 months of treatment; relapse: HCV-RNA that becomes positive again after treatment is stopped
* Compensated hepatic disease (Child-Pugh ≤ 6)
* Provision by patient of his or her written consent

Exclusion Criteria:

* Females who are pregnant or lactating will be excluded
* Renal failure (estimated glomerular filtration rate < 50 ml/min)
* A contraindication to treatment with peginterferon plus ribavirin (uncontrolled psychiatric illness, pregnancy/nursing/non-use of effective contraceptive method, uncontrolled epilepsy for at least 6 months, heart failure, unstable angina, hemoglobin < 120 g/L, neutrophils < 1,000/mm3, platelets < 50 x 109/L, or any other condition that, in the investigator's opinion, contraindicates use of the treatment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Hepatitis C Virus-Ribonucleic Acid (HCV-RNA) analysis assay | up to 24 weeks post treatment
  Qualitative

SECONDARY OUTCOMES:
Viral Kinetics | up to 24 weeks post treatment
  Plasma Ribavirin (RBV) Assays; Immune Response
Neutrophils | up to 24-48 weeks of treatment
  If neutrophils are < 500/mm, neupogen may be added
Hemoglobin | up to 24-48 weeks of treatment
  If hemoglobin is < 100g/L, erythropoietin and/or transfusions may be prescribed

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Villeneuve, M.D., Ph.D., Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Background] Tsubota A, Hirose Y, Izumi N, Kumada H. Pharmacokinetics of ribavirin in combined interferon-alpha 2b and ribavirin therapy for chronic hepatitis C virus infection. Br J Clin Pharmacol. 2003 Apr;55(4):360-7. doi: 10.1046/j.1365-2125.2003.01780.x. PMID 12680884
- [Background] Wade JR, Snoeck E, Duff F, Lamb M, Jorga K. Pharmacokinetics of ribavirin in patients with hepatitis C virus. Br J Clin Pharmacol. 2006 Dec;62(6):710-4. doi: 10.1111/j.1365-2125.2006.02704.x. PMID 17118126
- [Background] Maynard M, Pradat P, Gagnieu MC, Souvignet C, Trepo C. Prediction of sustained virological response by ribavirin plasma concentration at week 4 of therapy in hepatitis C virus genotype 1 patients. Antivir Ther. 2008;13(4):607-11. PMID 18672540
- [Background] Cheruvattath R, Rosati MJ, Gautam M, Vargas HE, Rakela J, Balan V. Pegylated interferon and ribavirin failures: is retreatment an option? Dig Dis Sci. 2007 Mar;52(3):732-6. doi: 10.1007/s10620-006-9457-x. PMID 17253142
- [Background] Glue P. The clinical pharmacology of ribavirin. Semin Liver Dis. 1999;19 Suppl 1:17-24. PMID 10349689
- [Background] Uchida M, Hamada A, Yamasaki M, Fujiyama S, Sasaki Y, Saito H. Assessment of adverse reactions and pharmacokinetics of ribavirin in combination with interferon alpha-2b in patients with chronic hepatitis C. Drug Metab Pharmacokinet. 2004 Dec;19(6):438-43. doi: 10.2133/dmpk.19.438. PMID 15681898
- [Background] Arase Y, Ikeda K, Tsubota A, Suzuki F, Suzuki Y, Saitoh S, Kobayashi M, Akuta N, Someya T, Hosaka T, Sezaki H, Kobayashi M, Kumada H. Significance of serum ribavirin concentration in combination therapy of interferon and ribavirin for chronic hepatitis C. Intervirology. 2005;48(2-3):138-44. doi: 10.1159/000081741. PMID 15812187
- [Background] Badr G, Bedard N, Abdel-Hakeem MS, Trautmann L, Willems B, Villeneuve JP, Haddad EK, Sekaly RP, Bruneau J, Shoukry NH. Early interferon therapy for hepatitis C virus infection rescues polyfunctional, long-lived CD8+ memory T cells. J Virol. 2008 Oct;82(20):10017-31. doi: 10.1128/JVI.01083-08. Epub 2008 Jul 30. PMID 18667516
- [Background] Hofer H, Donnerer J, Sator K, Staufer K, Scherzer TM, Dejaco C, Sator M, Kessler H, Ferenci P. Seminal fluid ribavirin level and functional semen parameters in patients with chronic hepatitis C on antiviral combination therapy. J Hepatol. 2010 Jun;52(6):812-6. doi: 10.1016/j.jhep.2009.12.039. Epub 2010 Mar 23. PMID 20399525
- [Background] Jen JF, Glue P, Gupta S, Zambas D, Hajian G. Population pharmacokinetic and pharmacodynamic analysis of ribavirin in patients with chronic hepatitis C. Ther Drug Monit. 2000 Oct;22(5):555-65. doi: 10.1097/00007691-200010000-00010. PMID 11034261
- [Background] Jen J, Laughlin M, Chung C, Heft S, Affrime MB, Gupta SK, Glue P, Hajian G. Ribavirin dosing in chronic hepatitis C: application of population pharmacokinetic-pharmacodynamic models. Clin Pharmacol Ther. 2002 Oct;72(4):349-61. doi: 10.1067/mcp.2002.127112. PMID 12386637
- [Background] Jensen DM, Marcellin P, Freilich B, Andreone P, Di Bisceglie A, Brandao-Mello CE, Reddy KR, Craxi A, Martin AO, Teuber G, Messinger D, Thommes JA, Tietz A. Re-treatment of patients with chronic hepatitis C who do not respond to peginterferon-alpha2b: a randomized trial. Ann Intern Med. 2009 Apr 21;150(8):528-40. doi: 10.7326/0003-4819-150-8-200904210-00007. PMID 19380853
- [Background] Kauppila A, Cantell K, Janne O, Kokko E, Vihko R. Serum sex steroid and peptide hormone concentrations, and endometrial estrogen and progestin receptor levels during administration of human leukocyte interferon. Int J Cancer. 1982 Mar 15;29(3):291-4. doi: 10.1002/ijc.2910290311. PMID 6175589
- [Background] Loustaud-Ratti V, Alain S, Rousseau A, Hubert IF, Sauvage FL, Marquet P, Denis F, Lunel F, Cales P, Lefebvre A, Fauchais AL, Liozon E, Vidal E. Ribavirin exposure after the first dose is predictive of sustained virological response in chronic hepatitis C. Hepatology. 2008 May;47(5):1453-61. doi: 10.1002/hep.22217. PMID 18435468
- [Background] Maeda Y, Kiribayashi Y, Moriya T, Maruhashi A, Omoda K, Funakoshi S, Murakami T, Takano M. Dosage adjustment of ribavirin based on renal function in Japanese patients with chronic hepatitis C. Ther Drug Monit. 2004 Feb;26(1):9-15. doi: 10.1097/00007691-200402000-00004. PMID 14749543